CLINICAL TRIAL: NCT06016205
Title: Ultrasound-guided PECS2 (The Pectoralis) Block Versus Intrathecal Morphine for Postoperative Analgesia After Mastectomy
Brief Title: The Pectoralis (PECS2) Block Versus Intrathecal Morphine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Mahmoud, Lecturer of anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Soh-Med-22-07-33
Record Dates: First submitted 2023-04-29; First posted 2023-08-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine group (n= 25): (Active Comparator)
  Interventions: Procedure: intrathecal morphine injection
- PECS group (n= 25): (Active Comparator)
  Interventions: Procedure: ultrasound guided PECS2 block

INTERVENTIONS:
Procedure: intrathecal morphine injection — Patients will receive intrathecal 200 microgram morphine immediately before induction of general anesthesia
  Arms: Morphine group (n= 25):
Procedure: ultrasound guided PECS2 block — ultrasound guided PECS2 block will be performed with 30 ml bupivacaine 0.25%
  Arms: PECS group (n= 25):

SUMMARY:
50 patients with American Society of Anesthesiologists (ASA) grade I to II, 18 to 60 years of age scheduled for Modified Radical Mastectomy surgery, Will be included in the study.

DETAILED DESCRIPTION:
Patients will be randomly divided into two groups:

morphine group (n=25):

Patients will receive intrathecal 200 microgram morphine immediately before induction of general anesthesia.

PECS group (n= 25):

PECS2 block will be performed and Patients will receive 30 ml bupivacaine 0.25% The drug solutions will be prepared by an anesthesiologist not involved in the study, the anesthesiologist performing the block and observing the patients will be blinded to the treatment group. Data collection will be done by anesthesiologist unaware of the group allocation.

In the PECS group patients will be placed in supine position. The block will be performed on the side of surgery with the ipsilateral upper limb in abduction position. After the skin of the infraclavicular region disinfected and preparing the US probe and adjusting the depth of 4 to 6cm and gain of Ultrasound machine .The 20-gauge echogenic needle will be introduced in-plane approach from medial to lateral and 10ml of bupivacaine 0.25% will be injected into the fascial plane between pectoralis muscles in order to block medial and lateral pectoral nerve (PECS I). Then the needle will be reinserted into the fascial plane between pectoralis minor and serratus anterior muscle and 20ml of bupivacaine 0.25%will be injected in increments of 5 ml after negative aspiration in order to block intercostals II-III-IV-V-VI and the long thoracic nerve.

General anesthesia will be induced in all patients with fentanyl (1-2ug/kg), propofol (1-2mg/kg) and an intuitive dose of atracurium (0. 5mg/kg), endotracheal intubation secured the airway. Anesthesia will be maintained with isoflurane (1- 2%) and an incremental dose of atracurium 0.1mg/kg. Controlled ventilation will be accomplished by a ventilator with a tidal volume of 6-8 ml/kg and an I/E ratio of 1:2 to maintain a tidal carbon dioxide voltage of approximately 35-40 mmHg.

The heart rate (HR), noninvasive arterial systolic blood pressure (SBP), diastolic blood pressure (DBP) and peripheral oxygen saturation (SpO2) will be recorded at baseline, after induction and with skin incision and every 5 minutes intraoperative till the end of surgery. And postoperative at 30 min, 1, 2, 3, 6, 12 and 24 hours.

- Postoperative pain will be assessed using visual analog score (VAS) [0-10]. 0 - 3 mild pain

* 4 - 6 moderate pain
* 7 - 10 severe pain
* 10 <unbearable pain)

All patients will receive paracetamol (1gm) immediately postoperative and every 6 hours. Patients will be assessed every one hour in the first 6 hours then every 4 hours in the next 18 hours. Patients will receive ketorolac 30 mg if VAS 3-5. If VAS>5, morphine 0.1mg/kg will be given then total ketorolac and morphine consumption in 24 hours will be calculated and compared between both groups.

Adverse effects will be considered as -bradycardia (if heart rate [HR] is <20% of baseline) will be treated by atropine (IV) 0.01 mg/kg.

* Hypotension (if mean arterial blood pressure is <20% of baseline) will be treated with (IV) fluid and an incremental (IV) dose of ephedrine 0.2- 0.3 mg/kg or (SC/IM) dose of ephedrine 0.5 mg/kg.
* Respiratory depression, apnea and hypoxemia (spo2 < 92%) will be treated with O2 supplementation.
* Also, complications as disturbed conscious level, nausea, vomiting and prolonged motor block will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) grade I to II, 18 to 60 years of age scheduled for Modified Radical Mastectomy surgery.

Exclusion Criteria:

* - Patient refusal.
* Patient with significant neurological , psychiatric or neuromuscular disease
* Alcoholism. Drug abuse.
* Pregnancy or lactating women.
* Suspected Coagulopathy.
* Morbid obesity.
* Known allergy to study medications.
* local infection at the block site

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
post-operative analgesia. | he visual analog score will be evaluated every 1 hour postoperatively.
  the visual analog score will be evaluated postoperatively in all the patients in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt